CLINICAL TRIAL: NCT03415958
Title: A Prospective Cohort of Displaced Adolescent Midshaft Clavicle Fractures: Are Times to Return to Activities and Functional Outcomes Reasonable for This Population?
Brief Title: A Prospective Cohort of Displaced Adolescent Midshaft Clavicle Fractures
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Edward Harvey, Orthopaedic Surgeon, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 10-358-PED
Record Dates: First submitted 2014-04-03; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Malunion of Fracture of Clavicle; Delayed Union of Fracture of Clavicle
Keywords: prospective; adolescent; displaced; clavicle; fracture; mid-shaft
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open reduction internal fixation: Patients with displaced midshaft clavicle fractures will be offered operative treatment which involves open reduction and internal fixation.
- Conservative care: Patients will be treated in a sling for the acute phase of two weeks with progressive physiotherapy.

SUMMARY:
Outcomes for displaced midshaft clavicle fractures in adolescents are not defined. The current method of treatment for these fractures is non-operative management. There is recent Level 1 evidence in the adult literature to suggest that outcomes are superior when these fractures are managed surgically with open reduction and internal fixation.

DETAILED DESCRIPTION:
The study is a prospective observational cohort design of the natural history of adolescent clavicle fractures treated at the McGill University Health Centre. Surgeon choice will dictate treatment. There is no difference from the current normal therapy choice of each individual surgeon. Patients will be offered either operative or conservative management.

Operative Treatment: Patients with displaced midshaft clavicle fractures will be offered operative treatment which involves open reduction and internal fixation with a plate. This is the standard treatment for completely displaced fractures in the adult population at our Institution based on Level 1 evidence.

Conservative care: Patients will be treated in a sling for the acute phase of two weeks with progressive physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-18 years old
* The only fracture present in that upper extremity
* Individual and/or parents able to comply with follow-up

Exclusion Criteria:

* Head injury
* Prior injury, degenerative condition or congenital condition of the upper extremities
* Systemic disease that may impair healing
* Incapable of ensuring follow-up

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents (ages 12 to 18) who have a displaced clavicle fracture
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2012-03-28 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Malunion and/or non-union in this cohort | 3 months
  Radiographic evaluation

SECONDARY OUTCOMES:
Times to union (clinical and radiographic) following fracture | 3 months
  Radiologic evaluation

OTHER OUTCOMES:
Visual Analogue Scale | 6 weeks, 3 months, 6 months, 12 months
  a measurement instrument for subjective characteristics which cannot be directly measured
Constant Shoulder Score | 6 weeks, 3 months, 6 months, 12 months
  a measurement instrument for strength, range of motion, power
Disabilities of the Arm, Shoulder and Hand | 6 weeks, 3 months, 6 months, 12 months
  a questionnaire
Activities & Your Injury | 6 weeks, 3 months, 6 months, 12 months
  a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Edward J. Harvey, MDCM, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Background] Vander Have KL, Perdue AM, Caird MS, Farley FA. Operative versus nonoperative treatment of midshaft clavicle fractures in adolescents. J Pediatr Orthop. 2010 Jun;30(4):307-12. doi: 10.1097/BPO.0b013e3181db3227. PMID 20502227
- [Background] Taylor DC, Krasinski KL. Adolescent shoulder injuries: consensus and controversies. J Bone Joint Surg Am. 2009 Feb;91(2):462-73. No abstract available. PMID 19181993
- [Background] Kocher MS, Waters PM, Micheli LJ. Upper extremity injuries in the paediatric athlete. Sports Med. 2000 Aug;30(2):117-35. doi: 10.2165/00007256-200030020-00005. PMID 10966151
- [Background] Hill JM, McGuire MH, Crosby LA. Closed treatment of displaced middle-third fractures of the clavicle gives poor results. J Bone Joint Surg Br. 1997 Jul;79(4):537-9. doi: 10.1302/0301-620x.79b4.7529. PMID 9250733
- [Background] McKee MD, Wild LM, Schemitsch EH. Midshaft malunions of the clavicle. J Bone Joint Surg Am. 2003 May;85(5):790-7. doi: 10.2106/00004623-200305000-00003. PMID 12728026
- [Background] McKee MD, Pedersen EM, Jones C, Stephen DJ, Kreder HJ, Schemitsch EH, Wild LM, Potter J. Deficits following nonoperative treatment of displaced midshaft clavicular fractures. J Bone Joint Surg Am. 2006 Jan;88(1):35-40. doi: 10.2106/JBJS.D.02795. PMID 16391247
- [Background] Ledger M, Leeks N, Ackland T, Wang A. Short malunions of the clavicle: an anatomic and functional study. J Shoulder Elbow Surg. 2005 Jul-Aug;14(4):349-54. doi: 10.1016/j.jse.2004.09.011. PMID 16015232
- [Background] McGraw MA, Mehlman CT, Lindsell CJ, Kirby CL. Postnatal growth of the clavicle: birth to 18 years of age. J Pediatr Orthop. 2009 Dec;29(8):937-43. doi: 10.1097/BPO.0b013e3181c11992. PMID 19934713
- [Background] Mehlman CT, Yihua G, Bochang C, Zhigang W. Operative treatment of completely displaced clavicle shaft fractures in children. J Pediatr Orthop. 2009 Dec;29(8):851-5. doi: 10.1097/BPO.0b013e3181c29c9c. PMID 19934697
- [Background] Zlowodzki M, Zelle BA, Cole PA, Jeray K, McKee MD; Evidence-Based Orthopaedic Trauma Working Group. Treatment of acute midshaft clavicle fractures: systematic review of 2144 fractures: on behalf of the Evidence-Based Orthopaedic Trauma Working Group. J Orthop Trauma. 2005 Aug;19(7):504-7. doi: 10.1097/01.bot.0000172287.44278.ef. PMID 16056089
- [Background] Canadian Orthopaedic Trauma Society. Nonoperative treatment compared with plate fixation of displaced midshaft clavicular fractures. A multicenter, randomized clinical trial. J Bone Joint Surg Am. 2007 Jan;89(1):1-10. doi: 10.2106/JBJS.F.00020. PMID 17200303